CLINICAL TRIAL: NCT04641117
Title: Time Efficient Exercise to Reverse Sarcopenia and Improve Cardio-metabolic Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTexasAustinKHE
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Exercise Training and Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Subjects will power train
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Six months of power training
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Walking and Power Training

SUMMARY:
Participants will be 60-80 y men and women who vary their physical activity (steps/day) while their lipid metabolism is studied (n=24). Thereafter, another group (n=60) will perform 6 months of exercise training focused on developing maximal cycling power, during which their changes in muscle mass and practical function will be carefully measured.

DETAILED DESCRIPTION:
In a society that is growing in the number of older adults who are also becoming more sedentary, it is critical to identify the types of exercise that harness significant health benefits. First, we hypothesize that older adults (60-80 y) need a certain background level of physical activity, judged by number of steps per day. This is important, especially to fat metabolism. Secondly, because older adults claim they don't have time to exercise, we have developed a time efficient program (10 min/day) that has shown promise for offsetting sarcopenia and significantly improving cardiovascular function.

Our Aim 1 is to determine the range of daily step counts in older adults (60-80 y; n=24) that is needed to prevent acute impairment of post-prandial fat metabolism, measured the morning after exercise. We have recently shown in young adults that when their level of background physical activity drops below the range of 5,000 - 8,500±500 steps/d, that they don't adapt positively to an acute 1 h bout of exercise (i.e.; 'exercise resistance') that normally improves fat metabolism.

Our Aim 2 is to determine the ability of a time-efficient 24-week program of exercise training for both maximal neuromuscular power and aerobic power to counteract sarcopenia and declines in aerobic power and functional tests in men and women 60-80 y. We have recently found in a preliminary study of older men and women (50-70 y) that performing multiple maximal 4 s sprints of rapid acceleration cycling bouts for only 8 weeks, eliciting maximal power, displayed significant (p<0.05) increases in muscle thigh volume (MRI), whole body muscle mass, maximal neuromuscular power and peak oxygen consumption. We now propose to train older men and women (i.e.; 60-80 y; n=60) for longer durations (i.e.; 24 weeks) and describe the time course of adaptations. We will additionally monitor their background levels of daily physical activity and determine if it correlates with improvements in neuromuscular and cardiovascular function.

ELIGIBILITY:
Inclusion Criteria:

* relatively healthy

Exclusion Criteria:

* relatively unhealthy

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle mass | six months
  MRI determined changes in thigh muscle volume
Post-prandial lipemia | one month
  The elevation of plasma triglycerides after a meal

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin Human Performance Laboratory, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No